CLINICAL TRIAL: NCT03105856
Title: HPV Vaccination Impact on Cervical Cancer Screening Program: FASTER-Tlalpan Study in Mexico
Brief Title: FASTER-Tlalpan Study in Mexico: HPV Vaccination Impact on Cervical Cancer Screening Program
Acronym: FASTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Principal Investigator, JORGE SALMERON, Principal Researcher, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1417
Record Dates: First submitted 2017-01-24; First posted 2017-04-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Cervical Intraepithelial Neoplasia; HPV-Related Cervical Carcinoma
Keywords: Mass screening; Vaccination; Mexico
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — human papillomavirus vaccine, L1 type 16, 18; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CERVARIX (Active Comparator): hrHPV-based screening and HPV16/18 L1 VLP AS04 vaccine (Cervarix®) group according to a two-dose schedule (0-12 months)
  Interventions: Biological: CERVARIX; Biological: GARDASIL
- GARDASIL (Active Comparator): hrHPV-based screening and Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) (Gardasil®) vaccine group according to a two-dose schedule (0-12 months)
  Interventions: Biological: CERVARIX; Biological: GARDASIL
- CONTROL GROUP (No Intervention): Control group who will receive only hrHPV-based screening.

INTERVENTIONS:
Biological: CERVARIX — - HPV16/18 L1 VLP AS04 vaccine (Cervarix®) group according to a two-dose schedule (0-12 month). This group will receive the HPV16/18 vaccine containing HPV16 and HPV18 L1 virus-like-particles (20 μg of each) adjuvanted with 50 μg 3-O-desacyl-4'-monophosphoryl lipid A and 0.5 mg aluminum hydroxide (GlaxoSmithKline Biologicals, Rixensart, Belgium). A 0.5-mL dose of the vaccine will be administered in the non-dominant arm.
  Arms: CERVARIX; GARDASIL
Biological: GARDASIL — Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) (Gardasil®) recombinant vaccine according to a two dose schedule (0-12 month). This group will receive amorphous aluminum hydroxyphosphate sulfate adjuvanted quadrivalent HPV (types 6, 11, 16, 18) L1 VLP vaccine (Merck Sharp & Dohme Corp. Whitehouse Station, NJ, USA). A 0.5-mL dose of the vaccine will be administered in the non-dominant arm.
  Arms: CERVARIX; GARDASIL

SUMMARY:
Objective. To evaluate the impact of HPV vaccination as part of a hrHPV-based primary screening program to extend screening intervals.

Materials and methods. A total of 3,000 women aged 25-45 years, attending the regular cervical cancer-screening program in primary health care services in Tlalpan, Mexico City, will be invited to the study. Eligible participants will be assigned to one of three comparison groups: 1) HPV16/18 vaccine and hrHPV-based screening; 2) HPV6/11/16/18 vaccine and hrHPV-based screening; 3) Control group who will receive only hrHPV-based screening. Strict surveillance of hrHPV persistent infection and occurrence of precancerous lesions will be conducted to estimate safety profiles at different screening intervals; participants will undergo diagnosis confirmation and treatment as necessary.

Discussion: The FASTER-Tlalpan Study will provide insights into new approaches of cervical cancer prevention programs. It will offer valuable information on potential benefits of combining HPV vaccination and hrHPV-based screening to safety extend screening intervals.

DETAILED DESCRIPTION:
Cervical cancer mortality is a reflection of social inequity in health care. Globally, 266,000 women die from cervical cancer annually, and 85% of these deaths occur in low- and middle income countries (LMIC).1,2 Persistent infection with high-risk human papillomavirus (hrHPV) is a necessary cause of cervical cancer.3,4 HPV16 and HPV18 are responsible for 70% of squamous cell carcinomas, and in conjunction with HPV45, cause 94.2% of cervical adenocarcinomas.4 The introduction of HPV vaccines will change the epidemiology of HPV-related cancers. However, it may take 30 years to observe the desired benefits of widespread vaccination when vaccinated cohorts reach the peak ages at which cervical cancer cases currently occur (e.g. women aged 40-50 years).5 As of August 2015, 84 countries and territories had national public-sector HPV immunization programs and 38 had pilot programs.6 These programs mainly target adolescent girls to obtain the greatest cost-benefit ratio,7 considering the initial price of the vaccine (>$100 US per dose).8,9 Women older than age 25 are also vulnerable to new HPV infections10 and could also be vaccinated depending on country-specific resource availability.

Recent results of Phase III HPV vaccination trials documented that the vaccine's efficacy among adult women is excellent (efficacy >80% to prevent resultant HPV-related cervical intraepithelial neoplasia).11,12 Additionally, current vaccines protect against both HPV16 and HPV18 as well as provide cross-protection against other HPV types, particularly types 31 and 45.13 Broad-spectrum protection such as this may lower the need for subsequent screening, warrant longer screening intervals than those currently used, and offer novel prevention policies against HPV-related cancers. The combination of vaccination and screening strategies to prevent cervical cancer may be particularly appropriate in countries with high incidence of cervical cancer that have already implemented hrHPV-based screening programs. These criteria are satisfied in Mexico.14 A broader age range of females in population-based HPV vaccination programs could have direct benefits for vaccinated females, and indirect benefits for non-vaccinated females and male sexual partners via increased herd immunity to reduce HPV-related cancers.15 Based on the high efficacy of the HPV vaccine in older women, a novel strategy combining vaccination and screening, HPV FASTER, has been proposed.16 In accordance with this proposal, HPV vaccination of women in a broad age range can offer protection to women who are not currently infected, but also can protect against subsequent re-infection.16 As a result, a combined strategy of HPV vaccination and screening may reduce the lifetime number of screens used by the current hrHPV-based screening programs. If a screening and vaccination strategy is widely adopted, we expect promising results. This strategy has the potential to: 1) mitigate the screening demand on both women and health services by extending screening intervals; 2) improve the cost-benefit balance of screening programs; and 3) provide greater protection and quality of life to a large number of women through a reduction in cervical cancer.17 An intervention such as this may not only save many lives in the next 30 years but also be cost-effective.

However, the data on efficacy of HPV vaccination in older women to reduce cervical cancer risk, and not just the risk of precancerous lesions, are lacking. That is, there is currently insufficient knowledge regarding the role of HPV vaccination in older women to permit screening intervals to be extend safely following a negative screen (Figure 1).

A significant challenge for HPV-vaccine uptake is the number of doses in the standard vaccine schedule. Although licensed in some countries for use among older individuals, national HPV vaccination programs target teenagers and young adults. Recent studies found that fewer than three doses of the two commercially available prophylactic HPV vaccines seem to provide similar protection against cervical HPV16 and HPV18 infections as the three-dose schedule in women younger than 25 years old. 18,19 Herein we propose a population-based study to assess the efficacy of a 2-dose HPV vaccination with [HPV16/18 AS04-adjuvanted vaccine (Cervarix ®) and HPV 6/11/16/18 vaccine (Gardasil®)] against HPV-persistent infection and HPV-related cervical disease in older women between 25 and 45 years of age attending clinics for hrHPV-based screening.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 25 to 45 years at the time of the first vaccine dose.
* Willing to comply with the requirements of the protocol (e.g., return for follow-up visits).
* Written informed consent prior to enrollment.

Exclusion Criteria:

* Pregnant or breastfeeding. Women must be at least 3 months post-pregnancy and not breastfeeding to enter the study.
* Planning to become pregnant or planning to discontinue contraceptive precautions during the first twelve months of the study (months 0-12).
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the vaccine.
* Any other medical condition or disease that could compromise the life of the participant during enrollment in the study.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days prior to the first dose of the study vaccine.
* Previous vaccination against human papillomavirus.
* History of cervical cancer or hysterectomy.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3000 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Inicidence 6-month persistent infection of HPV 16 or HPV 18 in women aged between 25-45 | During the study (10 years)
  The inicident 6-month persistent infection of HPV 16 or HPV 18 in women aged between 25-45 years, determining the positivity hrHPV with molecular techniques in orine samples after 30 and 36 months after a hrHPV-based screening after completion an average of 10 years of study

SECONDARY OUTCOMES:
Incidence of cervical intraepitelial neoplasia of grade 2 in women aged between 25-45 years | During the study (10 years)
  The incident of cervical intraepitelial neoplasia of grade 2 in women aged between 25-45 years, confirmed histologically by a biopsy after a positive hrHPV-based screening after completion an avarage of 10 years of study

CONTACTS AND LOCATIONS:
Overall Officials: JORGE SALMERON, PhD, Principal Investigator — Instituto Nacional de Salud Publica, Mexico
Locations (1):
- Jorge Salmeron, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Cancer Incidence and Mortality Worldwide: IARC CancerBase No. 11. International Agency for Research on Cancer. — http://globocan.iarc.fr.
- See also: ICO Information Centre on HPV and Cancer (HPV Information Centre). Human Papillomavirus and Related Diseases in the World. Summary Report. — http://www.hpvcentre.net/statistics/reports/XWX.pdf
- See also: Comisión Federal para la Protección contra Riesgos Sanitarios. Consulta de Registros Sanitarios 2015. — http://189.254.115.245/BuscadorPublicoRegistrosSanitarios/BusquedaRegistroSanitario.aspx